CLINICAL TRIAL: NCT03804645
Title: An Open-label, Randomized, Four-way Crossover Single Oral Dose Study Comparing the Pharmacokinetics of Four Different Formulations of AZD9977 (Part A) and Influence of Food and Lower Dose of a Selected Formulation (Part B) in Healthy Male Subjects
Brief Title: A Study to Assess the Reaction of Body for Four Different Formulations of AZD9977 (Part A) and Influence of Food and Lower Dose of a Selected Formulation (Part B) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6401C00006
Record Dates: First submitted 2019-01-14; First posted 2019-01-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
Keywords: Mineralocorticoid receptor; Heart failure with preserved ejection fraction; Safety; Pharmacokinetics; Influence of Food; Bioavailability
MeSH Terms: conditions — Heart Failure | interventions — AZD9977

STUDY DESIGN:
Intervention Model Description: open-label, randomized, four-way crossover single oral dose
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): In Part A, each subject will receive AZD9977 as a single dose on 4 different occasions under fasting conditions, separated by at least 48 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Cohort 2 (Experimental): In Part A, each subject will receive AZD9977 as a single dose on 4 different occasions under fasting conditions, separated by at least 48 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Cohort 3 (Experimental): In Part A, each subject will receive AZD9977 as a single dose on 4 different occasions under fasting conditions, separated by at least 48 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Cohort 4 (Experimental): In Part A, each subject will receive AZD9977 as a single dose on 4 different occasions under fasting conditions, separated by at least 48 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Cohort 5 (Experimental): In Part B, each subject will receive one formulation from Part A chosen for further development, dose under fed conditions, followed by dose under fasted condition.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D

INTERVENTIONS:
Drug: Treatment A — Each subject will receive single dose of AZD9977 capsule under fasting condition in Part A. If the formulation chosen for Part B, each subject will receive one dose under fed condition and another dose under fasted condition.
  Other Names: AZD9977 capsule, reference
Drug: Treatment B — Each subject will receive single dose of AZD9977 HDL capsule under fasting condition in Part A. If the formulation chosen for Part B, each subject will receive one dose under fed condition and another dose under fasted condition.
  Other Names: AZD9977 HDL capsule
Drug: Treatment C — Each subject will receive single dose of AZD9977 ODL capsule under fasting condition in Part A. If the formulation chosen for Part B, each subject will receive one dose under fed condition and other dose under fasted condition.
  Other Names: AZD9977 ODL capsule
Drug: Treatment D — Each subject will receive single dose of AZD9977 tablet under fasting condition in Part A. If the formulation chosen for Part B, each subject will receive one dose under fed condition and another dose under fasted condition.
  Other Names: AZD9977 tablet

SUMMARY:
AZD9977 is an oral, selective mineralocorticoid receptor (MR) modulator. AZD9977 is a partial antagonist and partial agonist in reporter gene assays and has a different interaction pattern with the MR compared to eplerenone.

This study will assess the pharmacokinetics (PK) of four different Formulations of AZD9977 (Part A) and influence of food and lower dose of a selected formulation (Part B) in healthy male subjects.

DETAILED DESCRIPTION:
This study will be a randomized, open-label, single-centre crossover study in healthy male subjects. The study is divided into 2 parts, Part A and Part B. The subjects will participate in both Part A and Part B.

Part A will be a 4-way cross-over study comparing the PK of AZD9977 as a reference capsule and 2 different capsule formulations and a tablet formulation under fasting conditions.

* Treatment A: Reference, AZD9977 capsule
* Treatment B: AZD9977 HDL capsule
* Treatment C: AZD9977 ODL capsule
* Treatment D: AZD9977 tablet In Part B, based on the interim results in Part A, 1 of the formulations will be selected and evaluated at the 300 mg dose level under fed conditions. The same formulation will also be evaluated under fasting conditions at a lower dose level (50 mg). The first dose tested in Part B will be the 50 mg (fasted) dose, followed by the 300 mg (fed) dose.

In Part A, subjects will be resident from 1 day before dosing (Day -1 of Treatment Period 1) with AZD9977 until 48 hours post-final-dose (Day 3 of Treatment Period 4). Subjects will return to the unit for Part B at least 48 hours (and up to 5 weeks) after completion of Part A.

In Part B, subjects will be resident from 1 day before dosing (Day -1 of Treatment Period 1) with AZD9977 until 48 hours post-final-dose (Day 3 of Treatment Period 2).

Subjects will return to the unit for a final study visit 5-7 days post-last-dose for a Follow up Visit.

Each subject will be involved in the study for approximately 12 weeks (including approximately 4 to 5 weeks for the interim analysis).

Twelve subjects will initially be randomized to ensure at least 8 and 6 evaluable subjects at the end of the last treatment period for Part A and Part B respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Agree to use the methods of contraception.
3. Healthy male subjects aged 18 to 50 years, inclusive, with suitable veins for cannulation or repeated venipuncture at screening.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive at screening.
5. Subject judged at screening likely to complete and agree to eat a specified high fat standardized Food and Drug Administration (FDA) breakfast.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the principal investigator (PI), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the PI, including:

   4.1. Serum potassium > 5.0 mmol/L.
5. Any clinically significant abnormal findings in vital signs, as judged by the PI, including:

   5.1. Systolic BP < 90 mmHg or > 140 mmHg. 5.2. Diastolic BP < 50 mmHg or > 90 mmHg. 5.3. Pulse rate < 45 or > 90 beats per minute.
6. Any clinically significant abnormalities on 12-lead echocardiogram (ECG), as judged by the PI.
7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
8. Known or suspected history of drug abuse in the 12 months prior to screening, as judged by the PI.
9. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of AZD9977 in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous Phase 1 study, are not excluded.
10. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977.
12. Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 3 months prior to screening.
13. Positive screen for drugs of abuse, alcohol or cotinine at screening or on admission to the study center.
14. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of AZD9977.
15. Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of AZD9977 or longer if the medication has a long half life.
16. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol in the 12 months prior to screening as judged by the PI.
17. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
18. Subjects who have previously received AZD9977.
19. Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
20. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUC) | At Dosing Session, For Part A (Days 1-3, 3-5, 5-7, 7-9) and For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To determine the relative bioavailability (Frel) and compare the plasma concentration time profile of 3 different formulations versus a reference capsule formulation of AZD9977 and to evaluate the influence of food by comparing AUC and Cmax under fasting and fed conditions for 1 of the formulations evaluated in Part A.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast) | At Dosing Session, For Part A (Days 1-3, 3-5, 5-7, 7-9) and For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To determine the relative bioavailability (Frel) and compare the plasma concentration time profile of 3 different formulations versus a reference capsule formulation of AZD9977 and to evaluate the PK of a lower dose of 1 of the formulations evaluated in Part A.
Area under the plasma concentration-time curve from time zero to 24 hours [AUC(0-24)] | At Dosing Session, For Part A (Days 1-3, 3-5, 5-7, 7-9) and For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To determine the relative bioavailability (Frel) and compare the plasma concentration time profile of 3 different formulations versus a reference capsule formulation of AZD9977 and to evaluate the PK of a lower dose of 1 of the formulations evaluated in Part A.
Maximum observed plasma concentration (Cmax) | At Dosing Session, For Part A (Days 1-3, 3-5, 5-7, 7-9) and For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To determine the relative bioavailability (Frel) and compare the plasma concentration time profile of 3 different formulations versus a reference capsule formulation of AZD9977 and to evaluate the influence of food by comparing AUC and Cmax under fasting and fed conditions for 1 of the formulations evaluated in Part A.
Observed AZD9977 concentration at 24 hours (C24) | At Dosing Session, For Part A (Days 1-3, 3-5, 5-7, 7-9) and For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To determine the relative bioavailability (Frel) and compare the plasma concentration time profile of 3 different formulations versus a reference capsule formulation of AZD9977 and to evaluate the PK of a lower dose of 1 of the formulations evaluated in Part A.
Area under plasma concentration-time curve from time zero to infinity divided by dose (AUC/D) | At Dosing Session, For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To evaluate the PK of a lower dose of 1 of the formulations evaluated in Part A.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration divided by dose (AUClast/D) | At Dosing Session, For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To evaluate the PK of a lower dose of 1 of the formulations evaluated in Part A
Area under the plasma concentration-time curve from time zero to 24 hours divided by dose [AUC(0-24)/D] | At Dosing Session, For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To evaluate the PK of a lower dose of 1 of the formulations evaluated in Part A
Maximum observed plasma concentration divided by dose (Cmax/D) | At Dosing Session, For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To evaluate the PK of a lower dose of 1 of the formulations evaluated in Part A
Observed AZD9977 concentration at 24 hours divided by dose (C24/D) | At Dosing Session, For Part B (Days 1-2, 3-4): Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post dose of each treatment
  To evaluate the PK of a lower dose of 1 of the formulations evaluated in Part A

SECONDARY OUTCOMES:
Number of subjects with Adverse events (AEs) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects
Number of subjects with abnormal blood pressure (BP) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects. Blood pressure includes both systolic and diastolic BP.
Number of subjects with abnormal pulse rate | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal findings in Real-Time Electrocardiogram (Cardiac Telemetry) | From Day-1 to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal findings in 12-lead safety Electrocardiogram (ECG) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal findings in physical examination | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects. The complete physical examinations will include the general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Number of subjects with abnormal laboratory assessments: absolute count of Basophils, Eosinophils, Monocytes, Neutrophils, Lymphocytes and Reticulocytes; Platelets and White blood cell (WBC) count | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Hematology- Red blood cell (RBC) count | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Hematology- Hemoglobin (Hb) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Hematology- Hematocrit (HCT) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects
Number of subjects with abnormal laboratory assessments: Hematology- Mean corpuscular volume (MCV) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Hematology- Mean corpuscular hemoglobin (MCH) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Hematology- Mean corpuscular hemoglobin concentration (MCHC) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry-Sodium | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry-Potassium | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Urea | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Creatinine | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Albumin | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Calcium | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Phosphate | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Glucose (fasting) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- C-reactive protein (CRP) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Alkaline phosphatase (ALP) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Alanine aminotransferase (ALT) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Aspartate aminotransferase (AST) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Gamma glutamyl transpeptidase (GGT) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Total Bilirubin (TBL) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Unconjugated bilirubin | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- High-sensitivity troponin T (hsTnT) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- Creatine kinase | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Serum Clinical Chemistry- N-terminal-pro-brain natriuretic peptide (NT-proBNP) | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Urinalysis-Glucose | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects.
Number of subjects with abnormal laboratory assessments: Urinalysis-Blood | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects. Microscopy will also be assessed if positive for blood): RBC count, WBC count, Casts (Cellular, Granular, Hyaline)
Number of subjects with abnormal laboratory assessments: Urinalysis-Protein | From screening (Day -28) to follow-up (Week 12)
  To assess the safety and tolerability of AZD9977 following oral administration in healthy male subjects. Microscopy will also be assessed if positive for protein): RBC count, WBC count, Casts (Cellular, Granular, Hyaline)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Forte Soto, MD, MSc, PhD, Principal Investigator — Dr.
Locations (1):
- Research Site, Harrow, United Kingdom

REFERENCES:
- See also: Study Information posted to AstraZeneca Cinical Trials Webiste — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/View?id=25801